CLINICAL TRIAL: NCT06664489
Title: Assessment of Knowledge, Attitude, and Practice of Primary Care Physicians Regarding Common Dermatologic Conditions in Sudan 2024: A Cross Sectional Study
Brief Title: Assessment of Knowledge, Attitude and Practice of Primary Care Doctors Towards Common Dermatologic Conditions in Sudan
Status: Completed | Type: Observational
Sponsor: Afifa Muhammad Alameen Khalifa Alshaykh (Other)
Responsible Party: Sponsor-Investigator, Afifa Muhammad Alameen Khalifa Alshaykh, Medicine Group Leader, Research and Publication office
Organization: Research and Publication office (Other)
Other Study IDs: 24003
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dermatological Disorders
Keywords: Dermatological conditions; skin disorders; Attitude; Knowledge; Primary care physicians; Sudan
MeSH Terms: conditions — Skin Diseases; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the knowledge, attitude, and practice of primary care physicians regarding the common dermatologic conditions in Sudan. The main question it aims to answer is:

What is the level of knowledge of primary healthcare doctors regarding common dermatological conditions in Sudan? what is the attitude and practice of primary healthcare doctors regarding common dermatological conditions in Sudan?

DETAILED DESCRIPTION:
Dermatological conditions represent a major global health burden and significant portion of primary healthcare visits. Primary healthcare physicians are the backbone of medical care and they are usually the first responders to deal with skin diseases. Therefore, it is essential for primary care doctors to possess the sufficient knowledge and the best practice to achieve the best possible outcomes. Assessing the knowledge, attitude and practice of doctors will help identify the areas of weakness and address the gaps.

Our online based cross-sectional study involved primary healthcare doctors across the 18 states of Sudan. The study utilized multistage sampling to select the participants to fill the online questionnaire that is intended to assess the knowledge of the participants using a photo quiz, the attitude using likert's scale based assessment and the practice.

the study explored the factors which may affect the knowledge attitude and practice of doctors like the age, sex, years of clinical experience, and number of cases seen per day.

ELIGIBILITY:
Inclusion Criteria:

* Primary care doctors above 23 years of age
* Work in primary healthcare settings in Sudan during the period of the study.

Exclusion Criteria:

* Doctors less than 23 years of age
* Not located in Sudan
* Didn't work in primary care facilities

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary healthcare doctors working in primary care facilities in Sudan
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Level of knowledge of common dermatological conditions in Sudan | April 2024 - September 2024
  The knowledge assessment quiz is scored out of 25 points, scores more than 60% of the correct answers is considered sufficient.
Attitude of primary healthcare doctors regarding common dermatological conditions in Sudan | April 2024 - September 2024
  five points likert-scale, 5 for strongly agree, 4 for agree, 3 for neutral, 2 for disagree, and 1 for strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- Research and Publication Office, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT06664489/Prot_SAP_000.pdf